CLINICAL TRIAL: NCT04224350
Title: Multi Center Randomized Open-label Phase IV Study to Compare the Efficacy and Safety After Conversion to TacroBell SR Capsule or TacroBell Capsule in Renal Transplant Patients Undergoing Maintenance Therapy With Reference Tacrolimus
Brief Title: Study to Evaluate the Efficacy and Safety of Tacrolimus in Kidney Transplant Recipients (BLOSSOM)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 211KT18017
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Kidney Transplant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Once-Daily Tacrolimus (Experimental): Experimental arm: TacroBell SR Cap.
  Interventions: Drug: TacroBell SR cap.
- Twice a Day Tacrolimus (Active Comparator): Active Comparator arm: TacroBell Cap.
  Interventions: Drug: Tacrolimus cap.

INTERVENTIONS:
Drug: TacroBell SR cap. — * Orally, once-daily in the morning
  * After first dose 0.2mg/kg, check the blood concentration of tacrolimus at each visit and adjust the dose to achieve the blood concentration maintaining at 3~12ng/ml for 0 to 3months and then at 3~8ng/ml for 3 to 6months of study treatment.
  Other Names: Tacrolimus SR cap.
  Arms: Once-Daily Tacrolimus
Drug: Tacrolimus cap. — * Orally, twice a day in the morning and night
  * After first dose 0.1mg/kg, check the blood concentration of tacrolimus at each visit and adjust the dose to achieve the blood concentration maintaining at 7~12ng/ml for 0 to 3months and then at 5~8ng/ml for 3 to 6months of study treatment.
  Arms: Twice a Day Tacrolimus

SUMMARY:
The purpose of this study is to evaluate the efficacy and Safety after conversion to TacroBell SR cap. or TacroBell cap. in patients who in renal transplant patients undergoing maintenance therapy with Reference Tacrolimus.

DETAILED DESCRIPTION:
This study is a multi-center, Randomized, Open-label and phase IV clinical trial that evaluates the efficacy and safety after conversion to TacroBell SR cap. or TacroBell cap. administration for 24 weeks in renal transplant patients undergoing maintenance therapy with Reference Tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

* Over 20 years old(male or female)
* Patients with eGFR (By CKD-EPI) ≥30mL/min/1.73m^2 and spot urine P/C ratio≤0.5 at screening test
* Patients who are taking Tacrolimus twice a day for maintenance therapy and have Trough level of 3~10ng/ml
* Agreement with written informed consent

Exclusion Criteria:

* Patients who have transplanted organs other than kidney
* Patients with acute rejection who have been clinically treated within the last month
* Patients who have changed their administration of adjuvant immunosuppressants and corticosteroids within the last month (dose change, discontinuation, etc.)
* Patients who have been diagnosed with cancer within the last 5 years (except skin cancer or thyroid cancer determined by the investigator that treatment has been completed)
* Patients deemed inappropriate for screening due to severe digestive disorders at screening
* Patients with severe systemic infections requiring treatment (transplantation may be possible after the infection is completely lost or controlled)
* Patients with genetic problems of galactose-intolerance, Lapp lactose deficiency or glucose-galactose malabsorption
* If the following cases occur during screening
* Treatment of active liver disease or increased one or more of the liver function tests (T-bilirubin, AST, ALT) levels more than three times the upper limit of normal range
* Patients with WBC <2,500/mm^3, PLT <75,000/mm^3, ANC <1,300/μL
* Patients who have experienced hypersensitivity reactions or serious abnormalities with medicines used in this clinical trial or with similar chemical structures (Tacrolimus, etc.)
* Pregnant or lactating women
* Patients of childbearing potential who do not agree to the proper use of contraception during the trial
* Patients who received other investigational drugs within 4 weeks prior to consent of the document
* Patients unable to participate in the clinical trial due to the judgment of other investigators

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite efficacy failure (biopsy-confirmed acute rejection; TCMR, graft loss, death, or follow-up failure) | until 24 weeks

SECONDARY OUTCOMES:
Incidence of biopsy-confirmed acute rejection(TCMR, AMR) | until 24 weeks
Pathologic Results, Occurrence, Treatment Methods, and Results of Acute Rejection Confirmed by Biopsy | until 24 weeks
Survival rate of transplanted organ | until 24 weeks
Survival rate of Patients | until 24 weeks
Serum-Cr value | until 24 weeks
eGFR(eGFR using CKD-EPI method) value | until 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Seoul, St.Mary's Hospital., Seoul, South Korea